CLINICAL TRIAL: NCT00840450
Title: Phase II Study of Paclitaxel With Imatinib Mesylate (Gleevec) in Taxane-pretreated Ovarian and Other Cancers of Mullerian Origin
Brief Title: Imatinib Mesylate (Gleevec) and Paclitaxel in Recurrent Patients of Ovarian and Other Cancers of Mullerian Origin
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: NYU Langone Health (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-226; CSTI57BUS224 (Other: Novartis)
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; recurrent; Gleevec; Paclitaxel; Taxane; mullerian
MeSH Terms: conditions — Ovarian Neoplasms; Recurrence | interventions — Imatinib Mesylate; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Paclitaxel + Imatinib Mesylate (Gleevec) (Experimental)
  Interventions: Drug: Gleevec/Paclitaxel

INTERVENTIONS:
Drug: Gleevec/Paclitaxel — One treatment cycle:
  Gleevec: 300 mg twice a day orally for 4 consecutive days, then off for 3 days, every 7 days for 28 days.
  Paclitaxel: 80 mg/m^2/week intravenously, 3 weeks on, one week off, every 28 days.
  After 3 treatment cycles, decision made to continue or not with the combination based on tolerance and lack of progression.
  Other Names: Gleevec:Imatinib Mesylate; Paclitaxel: Taxol

SUMMARY:
This study is designed to determine whether the combination treatment of Paclitaxel and Gleevec on recurrent ovarian cancer patients or other cancers of mullerian origin will generate better clinical response than Paclitaxel alone.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age.
* Histologically documented diagnosis of epithelial carcinoma arising in the ovary, fallopian tube or peritoneum, of any stage or grade at diagnosis. *Patients must have received initial cytoreductive surgery and chemotherapy with at least one platinum based chemotherapy regimen.

  *Eligible platinum resistant patients will have failed no more than two additional non platinum cytotoxic regimens for their persistent or recurrent disease.
* Measurable disease.
* Performance status 0, 1, 2 (Eastern Cooperative Oncology Group) .
* Adequate end organ function, defined as the following: total bilirubin < 1.5 x upper limit of normal (ULN), SGOT and SGPT < 2.5 x UNL, creatinine < 1.5 x ULN, ANC > 1.0 x 10E9/L, platelets > 100 x 10E9/L.
* Written, voluntary informed consent.

Exclusion Criteria:

* Patient has received any other anticancer treatment within 21 days of first day of study drug dosing and shown recovery of any recent drug-induced neutropenia and thrombocytopenia.
* Patient has another primary malignancy that has required active intervention within 5 years, with the exception of basal cell skin cancer or a cervical carcinoma in situ.
* Patient with Grade III/IV cardiac problems as defined by the New York Heart Association Criteria (i.e., congestive heart failure, myocardial infarction within 6 months of study).
* Patient has a severe and/or uncontrolled medical disease (i.e., uncontrolled diabetes, chronic renal disease, or active uncontrolled infection).
* Patients on coumadin-derived anticoagulants.
* Patient with brain metastasis.
* Chronic liver disease, Hep B or C.
* Patient has a known diagnosis of human immunodeficiency virus (HIV) infection.
* Patient received chemotherapy within 3 weeks -unless the disease is rapidly progressing.
* Patient previously received radiotherapy to at least 25 % of the bone marrow.
* Patient had a major surgery within 2 weeks prior to study entry.
* Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
* Patient is on any drug that may interfere with Gleevec (e.g., Dilantin, Coumadin,or others on the list on page 33-37 of the protocol).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-04; Primary Completion 2010-04 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco M Muggia, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU cancer center, New York, New York, United States

REFERENCES:
- See also: publication for this trial — http://www.ncbi.nlm.nih.gov/pubmed/20944093

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 patients were enrolled into this study from April 2007 to August 2009 from New York University medical center and affiliated hospitals. Only 12 were evaluable since 2 patients never received treatment because of rapid symptomatic deterioration.
Period: Overall Study
Arm/Group | Paclitaxel and Imatinib Mesylate (Gleevec)
Started | 12
Completed | 9
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel and Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 61 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 12
Platinum Sensitivity [Number; unit: Participants]
  Resistant | 10
  Sensitive | 2

OUTCOME MEASURES:

1. Primary Outcome: the Best Overall Clinical Response
Description: This is defined as the percentage of participants who had either a complete response (CR) or a partial response (PR) as the best overall response according to Response Evaluation Criteria in Solid Tumors (RECIST) for measurable disease or CA-125 criteria for non-measurable disease. The response is evaluated at 12 weeks of treatment.
Time Frame: 12 weeks
Population: The analysis is based on the intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel and Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 12
percentage of participants | 33

2. Secondary Outcome: Progression-free-tolerance
Description: This is defined as the percentage of participants who continued on treatment with no progression at 12 weeks since the start of treatment.A patient will be considered to have progression-free-tolerance if she does not drop out due to toxicity and does not have disease progression or die by the completion of 12 weeks on treatment.
Time Frame: 12 weeks
Population: Based on intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel and Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 12
percentage of participants | 75

3. Secondary Outcome: Progression-free-survival at 12 Months
Description: This defined as the percentage of participants who had progression free survival at 12 months from the beginning of the treatment.
Time Frame: up to 12 months
Population: Based on intent-to-treat population.
Measure: Number; unit: percentage of participants
Arm/Group | Paclitaxel and Imatinib Mesylate (Gleevec)
Number analyzed (Participants) | 12
percentage of participants | 17

ADVERSE EVENTS:
Time Frame: treatment period (up to 5 months) plus 30 days after treatment or until the the adverse events have resolved or returned to pretreatment values or deemed irreversible.
Arm/Group | Paclitaxel and Imatinib Mesylate (Gleevec)
Serious Adverse Events (participants affected / at risk) | 3/12
Other Adverse Events (participants affected / at risk) | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel and Imatinib Mesylate (Gleevec) (N=12)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel and Imatinib Mesylate (Gleevec) (N=12)
Alopecia (General disorders) | 5
Anemia (Blood and lymphatic system disorders) | 11
Diarrhea (Gastrointestinal disorders) | 5
Edema (General disorders) | 2
Fatigue (General disorders) | 9
Headache (General disorders) | 1
Mucostitis (Gastrointestinal disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Nausea (Gastrointestinal disorders) | 10
Neuropathy (Nervous system disorders) | 7
Neutropenia (Blood and lymphatic system disorders) | 5
Palpitation (Cardiac disorders) | 4
Shortness of breath (Cardiac disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
skin toxicity (Skin and subcutaneous tissue disorders) | 2

LIMITATIONS AND CAVEATS:
Premature closure led to small numbers of subjects analyzed (12 out of 50 targeted accrual number).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes